CLINICAL TRIAL: NCT04169295
Title: Gynecologists' Feedback on Assisted Reproductive Technology (ART) Birth Rates: a Randomized Controlled Trial
Brief Title: Gynecologists' Feedback on ART-Birth Rates
Acronym: GAB-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: s62972
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): At the time of their fresh embryo transfer couples will receive a document with the following feedback: a photo of their transferred embryo, the number of cryopreserved embryos, the quality rating of the transferred embryo's, and couple's personalized IVF-prognosis
  Interventions: Other: Gynecologists' feedback on ART-Birth rates
- Control group (Sham Comparator): At the time of their fresh embryo transfer couples will receive a document with a photo of their transferred embryo(s) and the number of cryopreserved embryos.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Gynecologists' feedback on ART-Birth rates — At the time of their fresh embryo transfer couples will receive a document with the following feedback: a photo of their transferred embryo, the number of cryopreserved embryos, the quality rating of the transferred embryo's and couple's personalized IVF-prognosis (i.e. their chance on a live birth from the current IVF-cycle, including the transfer of fresh and if available cryopreserved embryos), calculated by entering eight background characteristics and five IVF-laboratory results into a prognostic model.
  Arms: Intervention group
Other: Control group — At the time of their fresh embryo transfer couples will receive a document with the following feedback: a photo of their transferred embryo and the number of cryopreserved embryos
  Arms: Control group

SUMMARY:
The investigators will examine the hypothesis that women who are given their personalized IVF-prognosis are less likely to overestimate their IVF-live birth rate, as compared to women who do not receive a personalized IVF-prognosis.

Control group: At the time of their fresh embryo transfer couples will receive a document with a photo of their transferred embryo(s) and the number of cryopreserved embryos.

Intervention group: At the time of their fresh embryo transfer couples will receive a document with the following feedback: a photo of their transferred embryo, the number of cryopreserved embryos, the quality rating of the transferred embryo's, and couple's personalized IVF-prognosis (i.e. their chance on a live birth from the current IVF-cycle, including the transfer of fresh and if available cryopreserved embryos, calculated by entering eight background characteristics and five IVF-laboratory results into a prognostic model).

DETAILED DESCRIPTION:
Primary outcome:

The proportion of women expecting their IVF-live birth rate to be double their calculated IVF-prognosis, directly after their fresh embryo transfer.

Secondary outcomes:

The proportion of men expecting their IVF-live birth rate to be double their calculated IVF-prognosis, directly after their fresh embryo transfer.

Women's and men's anxiety will be assessed with the reliable 'State-Anxiety Inventory, (STAI-state)' questionnaire, disseminated in coded paper-pencil format on the day of the fresh embryo transfer.

Patient's infertility-specific distress will be assessed with the reliable 'Infertility Distress Scale (IDS)' questionnaire, within two days of the conclusive pregnancy test after the transfer of the last (fresh or cryopreserved) embryo of the studied IVF-cycle.

ELIGIBILITY:
Inclusion Criteria:

* Couples treated with a 2nd-6th fresh cycle of IVF (every couple can only participate ones in this study).

Exclusion Criteria:

* Couples treated with:

  * Pre-implantation Genetic Testing (PGT)
  * donated oocytes, sperm or embryos
  * Spermatozoa obtained by testicular extraction
  * HIV-positive diagnosis
  * Embryo transfer on day 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
The proportion of women over-estimating their IVF-live birth rate | Patient's expected IVF-live birth rate will be assessed immediately after the fresh embryo transfer with a single question coded paper-pencil questionnaire.
  The proportion of women expecting their IVF-live birth rate to be double their calculated IVF-prognosis, directly after their fresh embryo transfer.

SECONDARY OUTCOMES:
The proportion of men over-estimating their IVF-live birth rate | Patient's expected IVF-live birth rate will be assessed immediately after the fresh embryo transfer with a single question coded paper-pencil questionnaire.
  The proportion of men expecting their IVF-live birth rate to be double their calculated IVF-prognosis, directly after their fresh embryo transfer.
Women's and men's anxiety | Anxious feelings immediately after the fresh embryo transfer are assessed with the coded paper-pencil State Trait Anxiety Inventory, state module (STAI-state; 20-80, the higher, the more anxious)
  Women's and men's anxiety will be assessed with the reliable STAI-state questionnaire, disseminated in coded paper-pencil format on the day of the fresh embryo transfer.
Women's and men's infertility-specific distress | Infertility specific distress within 2 days of the conclusive pregnancy test after the the last embryotransfer (fresh or cryo) assessed with the Infertility Distress Scale (IDS; 8-40; the higher the more infertility specific distress)
  Women's and men's infertility-specific distress will be assessed with the reliable 'Infertility Distress Scale (IDS)' questionnaire, disseminated via text message and online

OTHER OUTCOMES:
Live birth rate of the observed IVF-cycle | Within 12-months after the oocyte aspiration of the observed IVF-cycle
  Cumulative clinical live birth rates after all embryo transfers resulting from the oocyte aspiration of the observed IVF-cycle
IVF-delay | Within 12-months after the oocyte aspiration of the observed IVF-cycle
  Number of untreated cycles prior to the start of a new fresh IVF-cycle after the last negative pregnancy test of the observed IVF-cycle
IVF-discontinuation | Within 12-months after the oocyte aspiration of the observed IVF-cycle
  Whether or not a subsequent IVF-cycle was started within twelve months after the last negative pregnancy test of the observed IVF-cycle and while no medical censoring to discontinue

CONTACTS AND LOCATIONS:
Overall Officials: Karen Peeraer, Prof., Principal Investigator — Leuven University Fertilitycentre
Locations (1):
- Leuven University Fertility Center, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT04169295/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT04169295/ICF_001.pdf